CLINICAL TRIAL: NCT00049517
Title: A Phase III Trial in Adult Acute Myeloid Leukemia: Daunorubicin Dose-Intensification Prior to Risk-Allocated Autologous Stem Cell Transplantation
Brief Title: Combination Chemotherapy With or Without Monoclonal Antibody Therapy in Treating Patients With AML Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258113; U10CA021115 (NIH); E1900 (Other: Eastern Cooperative Oncology Group (ECOG))
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Leukemia
Keywords: acute myeloid leukemia; autologous transplantation; gemtuzumab ozogamicin
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — sargramostim; Busulfan; Cyclophosphamide; Cytarabine; Gemtuzumab; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Standard Daunorubicin Then Autologous HCT (Experimental): Induction: Patients receive standard-dose daunorubicin IV over 10-15 minutes on days 1-3 and cytarabine IV continuously on days 1-7. Patients may receive a second course of induction therapy if complete remission (CR) is not achieved after the first course.
  Consolidation/Transplant:
  Before initiating consolidation therapy, patients with CR were randomized to a standard or an investigational arm. All patients received 2 cycles of high-dose cytarabine therapy (3 g/m2 given IV over a 3-hour period every 12 hours every other day for a total of 6 doses), followed by sargramostim 250 μg/m2 until recovery of blood counts.
  The patients undergoing autologous hematopoietic cell transplantation (HCT) received intravenous busulfan 0.8 mg/kg every 6 hours for 16 doses (without pharmacokinetic sampling) followed by intravenous cyclophosphamide 60 mg/kg daily for 2 days.
  Interventions: Biological: sargramostim; Drug: busulfan; Drug: cyclophosphamide; Drug: cytarabine; Drug: Daunorubicin; Procedure: Autologous HCT
- High-dose Daunorubicin Then Autologous HCT (Experimental): Induction: Patients receive high-dose daunorubicin IV over 10-15 minutes on days 1-3 and cytarabine IV continuously on days 1-7. Patients may receive a second course of induction therapy if complete remission (CR) is not achieved after the first course.
  Consolidation/Transplant:
  Before initiating consolidation therapy, patients with CR were randomized to a standard or an investigational arm. All patients received 2 cycles of high-dose cytarabine therapy (3 g/m2 given IV over a 3-hour period every 12 hours every other day for a total of 6 doses), followed by sargramostim 250 μg/m2 until recovery of blood counts.
  The patients undergoing autologous hematopoietic cell transplantation (HCT) received intravenous busulfan 0.8 mg/kg every 6 hours for 16 doses (without pharmacokinetic sampling) followed by intravenous cyclophosphamide 60 mg/kg daily for 2 days.
  Interventions: Biological: sargramostim; Drug: busulfan; Drug: cyclophosphamide; Drug: cytarabine; Drug: Daunorubicin; Procedure: Autologous HCT
- Standard Daunorubicin Then GO/Autologous HCT (Experimental): Induction: Patients receive standard-dose daunorubicin IV over 10-15 minutes on days 1-3 and cytarabine IV continuously on days 1-7. Patients may receive a second course of induction therapy if complete remission (CR) is not achieved after the first course.
  Consolidation/Transplant:
  Before initiating consolidation therapy, patients with CR were randomized to a standard or an investigational arm. All patients received 2 cycles of high-dose cytarabine therapy (3 g/m2 given IV over a 3-hour period every 12 hours every other day for a total of 6 doses), followed by sargramostim 250 μg/m2 until recovery of blood counts. patients randomized to the investigational arm received a single dose of Gemtuzumab ozogamicin (GO) at 6 mg/m2 followed by sargramostim 250 μ/m2 until recovery of counts.
  The patients undergoing autologous HCT received intravenous busulfan 0.8 mg/kg every 6 hours for 16 doses followed by intravenous cyclophosphamide 60 mg/kg daily for 2 days.
  Interventions: Biological: sargramostim; Drug: busulfan; Drug: cyclophosphamide; Drug: cytarabine; Drug: gemtuzumab ozogamicin (GO); Drug: Daunorubicin; Procedure: Autologous HCT
- High-dose Daunorubicin Then GO/Autologous HCT (Experimental): Induction: Patients receive high-dose daunorubicin IV over 10-15 minutes on days 1-3 and cytarabine IV continuously on days 1-7. Patients may receive a second course of induction therapy if complete remission (CR) is not achieved after the first course.
  Consolidation/Transplant:
  Before initiating consolidation therapy, patients with CR were randomized to a standard or an investigational arm. All patients received 2 cycles of high-dose cytarabine therapy (3 g/m2 given IV over a 3-hour period every 12 hours every other day for a total of 6 doses), followed by sargramostim 250 μg/m2 until recovery of blood counts. patients randomized to the investigational arm received a single dose of Gemtuzumab ozogamicin (GO) at 6 mg/m2 followed by sargramostim 250 μ/m2 until recovery of counts.
  The patients undergoing autologous HCT received intravenous busulfan 0.8 mg/kg every 6 hours for 16 doses followed by intravenous cyclophosphamide 60 mg/kg daily for 2 days.
  Interventions: Biological: sargramostim; Drug: busulfan; Drug: cyclophosphamide; Drug: cytarabine; Drug: gemtuzumab ozogamicin (GO); Drug: Daunorubicin; Procedure: Autologous HCT
- Standard Daunorubicin Then Allogeneic HCT or no Consolidation (Active Comparator): Induction: Patients receive standard-dose daunorubicin IV over 10-15 minutes on days 1-3 and cytarabine IV continuously on days 1-7. Patients may receive a second course of induction therapy if complete remission (CR) is not achieved after the first course.
  Consolidation/Transplant:
  Patients without CR did not receive any consolidation treatment. Patients in CR with an unfavorable cytogenetic profile or an initial white blood cell count > 100,000/μL were to proceed to allogeneic HCT if they had a suitable human leukocyte antigen (HLA)-matched sibling donor available.
  Interventions: Drug: cytarabine; Drug: Daunorubicin; Procedure: Allogeneic HCT
- High-dose Daunorubicin Then Allogeneic HCT or no Consolidation (Experimental): Induction: Patients receive high-dose daunorubicin IV over 10-15 minutes on days 1-3 and cytarabine IV continuously on days 1-7. Patients may receive a second course of induction therapy if complete remission (CR) is not achieved after the first course.
  Consolidation/Transplant:
  Patients without CR did not receive any consolidation treatment. Patients in CR with an unfavorable cytogenetic profile or an initial white blood cell count > 100,000/μL were to proceed to allogeneic HCT if they had a suitable human leukocyte antigen (HLA)-matched sibling donor available.
  Interventions: Drug: cytarabine; Drug: Daunorubicin; Procedure: Allogeneic HCT

INTERVENTIONS:
Biological: sargramostim — Given IV or as an injection
  Other Names: Leukine
  Arms: High-dose Daunorubicin Then Autologous HCT; High-dose Daunorubicin Then GO/Autologous HCT; Standard Daunorubicin Then Autologous HCT; Standard Daunorubicin Then GO/Autologous HCT
Drug: busulfan — Given IV
  Other Names: Myleran
  Arms: High-dose Daunorubicin Then Autologous HCT; High-dose Daunorubicin Then GO/Autologous HCT; Standard Daunorubicin Then Autologous HCT; Standard Daunorubicin Then GO/Autologous HCT
Drug: cyclophosphamide — Given IV
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune; cytophosphane
  Arms: High-dose Daunorubicin Then Autologous HCT; High-dose Daunorubicin Then GO/Autologous HCT; Standard Daunorubicin Then Autologous HCT; Standard Daunorubicin Then GO/Autologous HCT
Drug: cytarabine — Given as a continuous infusion
  Other Names: cytosine arabinoside
Drug: gemtuzumab ozogamicin (GO) — Given IV
  Other Names: Mylotarg
  Arms: High-dose Daunorubicin Then GO/Autologous HCT; Standard Daunorubicin Then GO/Autologous HCT
Drug: Daunorubicin — Given intravenously daily for 3 days at a dose of either 45 or 90 mg/m2.
  Other Names: daunomycin; daunomycin cerubidine
Procedure: Autologous HCT — Autologous hematopoietic cell transplantation
  Other Names: Autologous hematopoietic cell transplantation
  Arms: High-dose Daunorubicin Then Autologous HCT; High-dose Daunorubicin Then GO/Autologous HCT; Standard Daunorubicin Then Autologous HCT; Standard Daunorubicin Then GO/Autologous HCT
Procedure: Allogeneic HCT — Allogeneic hematopoietic cell transplantation
  Other Names: Allogeneic hematopoietic cell transplantation
  Arms: High-dose Daunorubicin Then Allogeneic HCT or no Consolidation; Standard Daunorubicin Then Allogeneic HCT or no Consolidation

SUMMARY:
RATIONALE: Giving combination chemotherapy before a stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the transplanted stem cells. When the healthy stem cells are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. If the patient's stem cells are to be transplanted, the patient is also treated with a monoclonal antibody, such as gemtuzumab ozogamicin, to kill any remaining cancer cells or deliver cancer-killing substances to them without harming normal cells. It is not yet known whether combination chemotherapy is more effective with or without gemtuzumab ozogamicin followed by stem cell transplant in treating acute myeloid leukemia.

PURPOSE: This randomized phase III trial is studying combination chemotherapy, gemtuzumab ozogamicin, and stem cell transplant to see how well they work compared to combination chemotherapy and peripheral stem cell transplant alone in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare the overall survival (OS) between two induction regimens (standard versus dose intense daunorubicin and cytarabine) in patients with de novo AML.
* To compare disease-free survival (DFS) between two consolidation regimens.
* To compare overall survival between two consolidation regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to induction therapy (standard-dose daunorubicin vs high-dose daunorubicin).

* Induction therapy: Patients are randomized to 1 of 2 induction arms.

  * Standard: Patients receive standard-dose daunorubicin IV over 10-15 minutes on days 1-3 and cytarabine IV continuously on days 1-7.
  * High dose: Patients receive high-dose daunorubicin IV over 10-15 minutes on days 1-3 and cytarabine as in arm I.

Patients in both arms may receive a second course of induction therapy if complete remission (CR) is not achieved after the first course. The second course is administered as in arm I to all patients. Patients who don't achieve CR after 2 courses of induction therapy are removed from study.

Patients who achieve CR after induction therapy proceed to post-remission therapy with EITHER allogeneic transplantation only (on or off study) OR consolidation therapy and autologous transplantation (on study), according to risk status and donor status.

Patients who are considered at intermediate or high risk for relapse (unfavorable cytogenetics/high WBC) and have a suitable related donor undergo an allogeneic transplantation. Patients with intermediate-risk cytogenetics, WBC no greater than 100,000/mm^3, and appropriate donors have the option of undergoing allogeneic transplantation.

* Allogeneic transplantation: Within 1-3 months after recovery from induction therapy, patients receive busulfan IV every 6 hours on days -7 to -4 and cyclophosphamide IV over 4 hours on days -3 and -2. Allogeneic bone marrow or peripheral blood stem cells (PBSCs) are infused on day 0. Patients receive graft-vs-host disease (GVHD) prophylaxis comprising cyclosporine IV over 1-4 hours beginning on day -1 and then orally (when tolerated) twice daily until day 180. Alternatively, patients may receive tacrolimus IV over 24 hours beginning on day -1 and then orally twice daily until day 180. Patients also receive methotrexate IV on days 1, 3, 6, and 11.

Patients who do not meet the criteria for allogeneic transplantation (i.e., are favorable risk or do not have a matching related donor) or who opt not to undergo allogeneic transplantation proceed to consolidation therapy followed by randomization to 1 of 2 autologous transplantation arms.

* Consolidation therapy: Beginning 2-8 weeks after recovery from induction therapy, patients receive high-dose cytarabine IV over 3 hours every 12 hours on days 1, 3, and 5. A second course is administered 3 weeks after blood recovery. Patients receive filgrastim (G-CSF) subcutaneously (SC) daily for 4 days and then autologous PBSCs are harvested by leukapheresis.
* Autologous stem cell transplantation: Patients are randomized to 1 of 2 autologous transplantation arms.

  * Arm I: Within 1 month after PBSC collection, patients receive conditioning comprising busulfan IV every 6 hours on days -7 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2. Patients then undergo autologous PBSC transplantation on day 0. Patients receive sargramostim (GM-CSF) or G-CSF IV or SC beginning on day 0 and continuing until blood counts recover.
  * Arm II (closed to accrual as of 10/4/2007): Within 2-4 weeks after PBSC collection, patients receive gemtuzumab ozogamicin IV over 2 hours on day 1 and GM-CSF SC or IV beginning on day 10 and continuing until blood counts recover. Within 2-3 weeks after blood count recovery, patients receive conditioning and undergo autologous PBSC transplantation as in arm I.

Patients are followed monthly for 1 year, every 2 months for 1 year, and then every 3 months for up to 7 years.

ACTUAL ACCRUAL: A total of 657 patients were accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Morphologically confirmed acute myeloid leukemia (AML) (greater than 20% blasts in the peripheral blood or marrow) meeting any of the following criteria:

  * Recurrent cytogenetic translocations

    * t(8;21)(q22;q22)
    * Bone marrow eosinophil abnormalities

      * inv(16)(p13;q22)
      * t(16;16)(p13;q22)
    * 11q23 abnormalities
  * Multilineage dysplasia without presence of myelodysplastic syndromes (MDS)
  * Minimally differentiated AML
  * AML without maturation
  * AML with maturation
  * AML not otherwise categorized
  * Acute myelomonocytic leukemia
  * Acute monocytic leukemia
  * Acute erythroid leukemia
  * Acute megakaryocytic leukemia
  * Acute basophilic leukemia
* Patients undergoing allogeneic transplantation must have a sibling donor match defined as human leukocyte antigen (HLA) match or haplotype match with one locus mismatch on other haplotype
* Age 16 to 60
* Eastern Cooperative Oncology Group (ECOG) performance status 0-4
* Aspartate aminotransferase (AST) less than 4 times upper limit of normal (ULN)
* Alkaline phosphatase less than 4 times ULN
* Creatinine no greater than 2.0 mg/dL
* Creatinine clearance at least 50 mL/min
* Left ventricular ejection fraction (LVEF) at least 45% by post-induction multigated acquisition (MUGA) scan
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* Prior hydroxyurea allowed
* Prior corticosteroids allowed

Exclusion Criteria:

* Recurrent cytogenetic translocations

  * Acute promyelocytic leukemia (PML) with t(15;17)(q22;q21)
  * Variant acute PML with t(v;17)
* Multilineage dysplasia with prior MDS
* Acute panmyelosis with myelofibrosis

  * Blastic transformation of chronic myelogenous leukemia
  * Secondary AML (chemotherapy-induced or evolved from MDS)
  * Pregnant or nursing
  * Bilirubin greater than 2.0 mg/dL (unless related to Gilbert's syndrome or hemolysis)
  * Significant cardiac disease requiring active therapy (e.g., digoxin, diuretics, antiarrhythmics, or antianginal medications)
  * Prior biologic therapy
  * Prior cytotoxic chemotherapy for any malignancy
  * Prior radiotherapy for any malignancy

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 657 (Actual)
Dates: Start 2002-12-19 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugo F. Fernandez, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (99):
- United States (98):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital - West, Boca Raton, Florida
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital - Main Campus, Boca Raton, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - La Grange Oncology Associates - Geneva, Naperville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Jewish Hospital Cancer Center, Cincinnati, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Rambam Medical Center, Haifa, Israel

REFERENCES:
- [Result] Fernandez HF, Sun Z, Yao X, Litzow MR, Luger SM, Paietta EM, Racevskis J, Dewald GW, Ketterling RP, Bennett JM, Rowe JM, Lazarus HM, Tallman MS. Anthracycline dose intensification in acute myeloid leukemia. N Engl J Med. 2009 Sep 24;361(13):1249-59. doi: 10.1056/NEJMoa0904544. PMID 19776406
- [Result] Fernandez HF, Sun Z, Bennett JM, et al.: A single dose of gemtuzumab-ozogamicin (GO) in consolidation prior to autologous transplant for younger patients with newly diagnosed acute myeloid (AML) is safe but has no effect on disease free survival: interim results of Eastern Cooperative Oncology Group study (E1900). [Abstract] Biol Blood Marrow Transplant 14 (2): A-52, 21-2, 2008.
- [Result] Vance GH, Kim H, Hicks GA, Cherry AM, Higgins R, Hulshizer RL, Tallman MS, Fernandez HF, Dewald GW. Utility of interphase FISH to stratify patients into cytogenetic risk categories at diagnosis of AML in an Eastern Cooperative Oncology Group (ECOG) clinical trial (E1900). Leuk Res. 2007 May;31(5):605-9. doi: 10.1016/j.leukres.2006.07.026. Epub 2006 Sep 22. PMID 16996130
- [Result] Fernandez HF, Kim HT, Bennett JM, et al.: Gemtuzumab-ozogamicin (GO; mylotarg®) as part of consolidation therapy for AML before autograft: low incidence of hepatic veno-occlusive disease. [Abstract] Biol Blood Marrow Transplant 11 (2 Suppl 1): A-187, 2005.
- [Result] Gonen M, Sun Z, Figueroa ME, Patel JP, Abdel-Wahab O, Racevskis J, Ketterling RP, Fernandez H, Rowe JM, Tallman MS, Melnick A, Levine RL, Paietta E. CD25 expression status improves prognostic risk classification in AML independent of established biomarkers: ECOG phase 3 trial, E1900. Blood. 2012 Sep 13;120(11):2297-306. doi: 10.1182/blood-2012-02-414425. Epub 2012 Aug 1. PMID 22855599
- [Result] Fernandez HF, Sun Z, Litzow MR, Luger SM, Paietta EM, Racevskis J, Dewald G, Ketterling RP, Rowe JM, Lazarus HM, Tallman MS. Autologous transplantation gives encouraging results for young adults with favorable-risk acute myeloid leukemia, but is not improved with gemtuzumab ozogamicin. Blood. 2011 May 19;117(20):5306-13. doi: 10.1182/blood-2010-09-309229. Epub 2011 Mar 17. PMID 21415269
- [Derived] Zarnegar-Lumley S, Alonzo TA, Gerbing RB, Othus M, Sun Z, Ries RE, Wang J, Leonti A, Kutny MA, Ostronoff F, Radich JP, Appelbaum FR, Pogosova-Agadjanyan EL, O'Dwyer K, Tallman MS, Litzow M, Atallah E, Cooper TM, Aplenc RA, Abdel-Wahab O, Gamis AS, Luger S, Erba H, Levine R, Kolb EA, Stirewalt DL, Meshinchi S, Tarlock K. Characteristics and prognostic impact of IDH mutations in AML: a COG, SWOG, and ECOG analysis. Blood Adv. 2023 Oct 10;7(19):5941-5953. doi: 10.1182/bloodadvances.2022008282. PMID 37267439
- [Derived] Foran JM, Sun Z, Lai C, Fernandez HF, Cripe LD, Ketterling RP, Racevskis J, Luger SM, Paietta E, Lazarus HM, Zhang Y, Bennett JM, Levine RL, Rowe JM, Litzow MR, Tallman MS. Obesity in adult acute myeloid leukemia is not associated with inferior response or survival even when dose capping anthracyclines: An ECOG-ACRIN analysis. Cancer. 2023 Aug 15;129(16):2479-2490. doi: 10.1002/cncr.34807. Epub 2023 Apr 25. PMID 37185873
- [Derived] Ganzel C, Sun Z, Baslan T, Zhang Y, Gonen M, Abdel-Wahab OI, Racevskis J, Garrett-Bakelman F, Lowe SW, Fernandez HF, Ketterling R, Luger SM, Litzow M, Lazarus HM, Rowe JM, Tallman MS, Levine RL, Paietta E. Measurable residual disease by flow cytometry in acute myeloid leukemia is prognostic, independent of genomic profiling. Leuk Res. 2022 Dec;123:106971. doi: 10.1016/j.leukres.2022.106971. Epub 2022 Oct 21. PMID 36332294
- [Derived] Luskin MR, Gimotty PA, Smith C, Loren AW, Figueroa ME, Harrison J, Sun Z, Tallman MS, Paietta EM, Litzow MR, Melnick AM, Levine RL, Fernandez HF, Luger SM, Carroll M, Master SR, Wertheim GB. A clinical measure of DNA methylation predicts outcome in de novo acute myeloid leukemia. JCI Insight. 2016 Jun 16;1(9):e87323. doi: 10.1172/jci.insight.87323. PMID 27446991
- [Derived] Luskin MR, Lee JW, Fernandez HF, Abdel-Wahab O, Bennett JM, Ketterling RP, Lazarus HM, Levine RL, Litzow MR, Paietta EM, Patel JP, Racevskis J, Rowe JM, Tallman MS, Sun Z, Luger SM. Benefit of high-dose daunorubicin in AML induction extends across cytogenetic and molecular groups. Blood. 2016 Mar 24;127(12):1551-8. doi: 10.1182/blood-2015-07-657403. Epub 2016 Jan 11. PMID 26755712
- [Derived] Walter RB, Othus M, Paietta EM, Racevskis J, Fernandez HF, Lee JW, Sun Z, Tallman MS, Patel J, Gonen M, Abdel-Wahab O, Levine RL, Estey EH. Effect of genetic profiling on prediction of therapeutic resistance and survival in adult acute myeloid leukemia. Leukemia. 2015 Oct;29(10):2104-7. doi: 10.1038/leu.2015.76. Epub 2015 Mar 16. No abstract available. PMID 25772026
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From December 19, 2002 through November 2008, a total of 657 patients were enrolled in the study.
Period: Induction
Arm/Group | Standard Daunorubicin Then Autologous HCT | High-dose Daunorubicin Then Autologous HCT | Standard Daunorubicin Then GO/Autologous HCT | High-dose Daunorubicin Then GO/Autologous HCT | Standard Daunorubicin Then Allogeneic HCT or no Consolidation | High-dose Daunorubicin Then Allogeneic HCT or no Consolidation
Started | 79 | 90 | 63 | 75 | 188 | 162
Treated | 79 | 90 | 63 | 75 | 186 | 160
Completed | 79 | 90 | 63 | 75 | 128 | 108
Not Completed | 0 | 0 | 0 | 0 | 60 | 54
Not completed — Disease progression | 0 | 0 | 0 | 0 | 18 | 11
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 5 | 7
Not completed — Death | 0 | 0 | 0 | 0 | 9 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Alternative therapy | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Other complicating disease | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Reasons not reported | 0 | 0 | 0 | 0 | 22 | 25
Period: Conditioning/Transplant
Arm/Group | Standard Daunorubicin Then Autologous HCT | High-dose Daunorubicin Then Autologous HCT | Standard Daunorubicin Then GO/Autologous HCT | High-dose Daunorubicin Then GO/Autologous HCT | Standard Daunorubicin Then Allogeneic HCT or no Consolidation | High-dose Daunorubicin Then Allogeneic HCT or no Consolidation
Started | 79 | 90 | 63 | 75 | 21 | 24
Randomized to Autologous HCT +/- GO | 59 (Additional 20 patients received Autologous HCT without randomization.) | 73 (Additional 17 patients received Autologous HCT without randomization.) | 63 | 75 | 0 (These 21 patients received Allogeneic HCT without randomization.) | 0 (These 24 patients received Allogeneic HCT without randomization.)
Completed | 27 | 40 | 25 | 32 | 15 | 18
Not Completed | 52 | 50 | 38 | 43 | 6 | 6
Not completed — Disease progression | 14 | 6 | 10 | 6 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 4 | 8 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 8 | 4 | 7 | 0 | 0
Not completed — Alternative therapy | 4 | 4 | 2 | 1 | 1 | 0
Not completed — Other complicating disease | 2 | 0 | 0 | 4 | 0 | 1
Not completed — Reasons not reported | 25 | 31 | 18 | 15 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Standard Daunorubicin (Induction Therapy): Patients receive standard-dose daunorubicin IV over 10-15 minutes on days 1-3 and cytarabine IV continuously on days 1-7.
  Patients may receive a second course of induction therapy if complete remission (CR) is not achieved after the first course.
- High Dose Daunorubicin (Induction Therapy): Patients receive high-dose daunorubicin IV over 10-15 minutes on days 1-3 and cytarabine as in arm I. Patients may receive a second course of induction therapy if CR is not achieved after the first course. The second course is administered as in arm I.
- Total: Total of all reporting groups
Arm/Group | Standard Daunorubicin (Induction Therapy) | High Dose Daunorubicin (Induction Therapy) | Total
Number analyzed (Participants) | 330 | 327 | 657
Age, Continuous [Median (Full Range); unit: years] | 47 [17 to 60] | 48 [18 to 60] | 48 [17 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 164 | 322
  Male | 172 | 163 | 335

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (Induction Phase)
Description: Overall survival is defined as the time from randomization in the induction phase to death.
Time Frame: Assessed during the first 4 months, then at least every three months for 2 years. then every six months until 5 years after study entry and every 12 months thereafter.
Population: All randomized patients are included in the analysis (intention-to-treat).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Standard Daunorubicin: Induction: Patients receive standard-dose daunorubicin IV over 10-15 minutes on days 1-3 and cytarabine IV continuously on days 1-7. Patients may receive a second course of induction therapy if complete remission (CR) is not achieved after the first course. Patients with CR received consolidation treatment thereafter.
- High-dose Daunorubicin: Induction: Patients receive high-dose daunorubicin IV over 10-15 minutes on days 1-3 and cytarabine IV continuously on days 1-7. Patients may receive a second course of induction therapy if complete remission (CR) is not achieved after the first course. Patients with CR received consolidation treatment thereafter.
Arm/Group | Standard Daunorubicin | High-dose Daunorubicin
Number analyzed (Participants) | 330 | 327
months | 15.7 [12.7 to 19.0] | 23.7 [19.0 to 31.7]

2. Primary Outcome: Disease-free Survival (Consolidation Phase)
Description: Disease-free survival is defined from the time of the confirmation of a complete remission via biopsy to the relapse of the disease.
Time Frame: Assessed during the first 4 months, then at least every three months for 2 years. then every six months until five years after study entry, and every 12 months thereafter.
Population: Only 270 patients who were randomized in the consolidation phase are included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Autologous HCT; Go/Autologous HCT: Patients with CR in the induction phase were randomized to receive autologous HCT or GO/autologous HCT.
Arm/Group | Autologous HCT | Go/Autologous HCT
Number analyzed (Participants) | 132 | 138
Months | 15.0 [11.4 to 23.9] | 13.6 [10.7 to 18.4]

3. Secondary Outcome: Overall Survival (Consolidation Phase)
Description: Overall survival is defined as the time from randomization in the consolidation phase to death.
Time Frame: as for outcome 2
Population: Only 270 patients who were randomized in the consolidation phase are included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Autologous HCT | Go/Autologous HCT
Number analyzed (Participants) | 132 | 138
Months | 35.5 [24.2 to 51.7] | 27.9 [20.3 to 39.5]

ADVERSE EVENTS:
Time Frame: Assessed weekly while on treatment and for 30 days after the end of treatment.
Groups:
- Standard Daunorubicin (Induction Therapy): Induction: Patients receive standard-dose daunorubicin IV over 10-15 minutes on days 1-3 and cytarabine IV continuously on days 1-7. Patients may receive a second course of induction therapy if complete remission (CR) is not achieved after the first course.
  Conditioning/Transplant:
  Patients receive conditioning comprising busulfan IV every 6 hours on days -7 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2. Patients then undergo autologous peripheral blood stem cell (PBSC) transplantation on day 0. Patients receive sargramostim (GM-CSF) or filgrastim (G-CSF) IV or subcutaneously (SC) beginning on day 0 and continuing until blood counts recover.
- High Dose Daunorubicin (Induction Therapy): Induction: Patients receive high-dose daunorubicin IV over 10-15 minutes on days 1-3 and cytarabine as in arm I. Patients may receive a second course of induction therapy if CR is not achieved after the first course. The second course is administered as in arm I.
  Conditioning/Transplant:
  Patients receive gemtuzumab ozogamicin IV over 2 hours on day 1 and GM-CSF SC or IV beginning on day 10 and continuing until blood counts recover. Within 2-3 weeks after blood count recovery, patients receive conditioning and undergo autologous PBSC transplantation as in arm I.
Arm/Group | Standard Daunorubicin (Induction Therapy) | High Dose Daunorubicin (Induction Therapy)
Serious Adverse Events (participants affected / at risk) | 328/328 | 325/325
Other Adverse Events (participants affected / at risk) | 319/328 | 318/325
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Daunorubicin (Induction Therapy) (N=328) | High Dose Daunorubicin (Induction Therapy) (N=325)
Bone Marrow Cellularity (Musculoskeletal and connective tissue disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 257 | 251
Hemolysis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 320 | 323
Lymphopenia (Blood and lymphatic system disorders) | 3 | 4
Neutropenia (Blood and lymphatic system disorders) | 319 | 305
Thrombocytopenia (Blood and lymphatic system disorders) | 321 | 321
Transfusion platelets (Blood and lymphatic system disorders) | 199 | 206
Transfusion: PRBCS (Blood and lymphatic system disorders) | 197 | 191
Hematologic-other (Blood and lymphatic system disorders) | 1 | 0
VOD (General disorders) | 1 | 1
Sinus Tachycardia (Cardiac disorders) | 0 | 2
Supraventricular arrhythmias (Cardiac disorders) | 1 | 6
Ventricular arrthhmia (Cardiac disorders) | 1 | 2
Arrhythmia-other (Cardiac disorders) | 0 | 1
Acute Vascular leak syndrome (Cardiac disorders) | 0 | 1
Cardiac ischemia (Cardiac disorders) | 0 | 1
Edema (General disorders) | 1 | 0
Hypertension (Blood and lymphatic system disorders) | 5 | 2
Hypotension (Blood and lymphatic system disorders) | 9 | 12
Thrombosis (Blood and lymphatic system disorders) | 4 | 2
Fatigue (General disorders) | 18 | 19
Fever (General disorders) | 22 | 29
Weight gain (Blood and lymphatic system disorders) | 1 | 0
Weight loss (General disorders) | 1 | 3
DIC (Blood and lymphatic system disorders) | 5 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 17 | 16
Wound-infectious (Infections and infestations) | 2 | 1
Anorexia (Psychiatric disorders) | 26 | 32
Colitis (Gastrointestinal disorders) | 6 | 8
Diarrhea (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 4
Nausea (Gastrointestinal disorders) | 19 | 16
Stomatitis (Ear and labyrinth disorders) | 9 | 20
Typhlitis (Gastrointestinal disorders) | 6 | 9
Vomiting (Gastrointestinal disorders) | 7 | 8
Epistaxis (General disorders) | 8 | 10
Bilirubin Increased (Blood and lymphatic system disorders) | 13 | 15
Hypoalbuminemia (Blood and lymphatic system disorders) | 5 | 3
AST increased (Blood and lymphatic system disorders) | 3 | 4
ALT Increased (Blood and lymphatic system disorders) | 10 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 121 | 117
hyperglycemia (Metabolism and nutrition disorders) | 7 | 4
Hypokalemia (Blood and lymphatic system disorders) | 0 | 1
Dyspnea (General disorders) | 18 | 13
Cardiac-Left Ventricular Function (Cardiac disorders) | 0 | 4
Cardiac Troponin I (Cardiac disorders) | 1 | 0
Operative Injury of Vein/Artery (Injury, poisoning and procedural complications) | 1 | 0
Pericardial Effusion/Pericarditis (Cardiac disorders) | 2 | 0
Cardiac-other (Cardiac disorders) | 1 | 2
Rigors/chills (General disorders) | 0 | 1
Constitutional symptoms (General disorders) | 1 | 0
PTT (Investigations) | 1 | 0
Hand-Foot Reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Wound - non-infectious (Injury, poisoning and procedural complications) | 0 | 1
Skin- Other (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flashes (Vascular disorders) | 0 | 1
SIADH (Investigations) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 3
Proctitis (Gastrointestinal disorders) | 4 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 7 | 12
Diarrhea w/ prior colostomy (Gastrointestinal disorders) | 1 | 1
GI-other (Gastrointestinal disorders) | 1 | 3
Hemorrhage with Grade 3 or 4 Platelets (Injury, poisoning and procedural complications) | 30 | 36
Hemorrhage without Grade 3 or 4 Platelets (Injury, poisoning and procedural complications) | 0 | 1
CNS hemorrhage (Blood and lymphatic system disorders) | 2 | 1
Hematemesis (Gastrointestinal disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hemorrhage Associated with Surgery (Injury, poisoning and procedural complications) | 1 | 1
Melena/GI Bleeding (Gastrointestinal disorders) | 0 | 4
Petechiae (Blood and lymphatic system disorders) | 5 | 2
Rectal Bleeding (Gastrointestinal disorders) | 1 | 1
Vaginal Bleeding (Reproductive system and breast disorders) | 3 | 1
Hemorrhage-Other (Vascular disorders) | 1 | 1
Alkaline phosphatase increased (Investigations) | 1 | 6
Infection w/ Gr3-4 neutropenia (Infections and infestations) | 154 | 168
Catheter-Related Infection (Infections and infestations) | 1 | 4
Infection w/ unknown ANC (Infections and infestations) | 1 | 1
Infection w/o neutropenia (Infections and infestations) | 10 | 13
Infection- Other (Infections and infestations) | 1 | 1
Acidosis (Infections and infestations) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 3
Hypokalemia (Metabolism and nutrition disorders) | 11 | 9
Hyponatremia (Metabolism and nutrition disorders) | 6 | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint, Muscle, Bone-Other (Musculoskeletal and connective tissue disorders) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 3 | 5
Depressed Level of consciousness (Psychiatric disorders) | 0 | 2
Dizziness/Lightheadedness (Nervous system disorders) | 4 | 0
Hallucinations (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Anxiety/Agitation (Psychiatric disorders) | 2 | 2
Depression (Psychiatric disorders) | 0 | 2
Neuropathy-motor (Nervous system disorders) | 1 | 0
Neuropathy-sensory (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 1
Speech Impairment (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 6 | 0
Ocular-Other (Nervous system disorders) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Bone, pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Chest Pain (General disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rectal or Perirectal Pain (Gastrointestinal disorders) | 2 | 2
Pain-other (General disorders) | 5 | 4
ARDS (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 | 13
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 12 | 14
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Creatinine increased (Investigations) | 2 | 1
Renal Failure (Renal and urinary disorders) | 3 | 3
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Daunorubicin (Induction Therapy) (N=328) | High Dose Daunorubicin (Induction Therapy) (N=325)
Anemia (Blood and lymphatic system disorders) | 319 | 318
Leukopenia (Blood and lymphatic system disorders) | 281 | 267
Neutropenia (Blood and lymphatic system disorders) | 243 | 230
Thrombocytopenia (Blood and lymphatic system disorders) | 295 | 292
Nausea (General disorders) | 16 | 18
Fatigue (General disorders) | 11 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No